CLINICAL TRIAL: NCT04223284
Title: Olfactory Odour Stimulation for Metabolism Control - the "OLFAMET-Study"
Brief Title: Olfactory Odour Stimulation for Metabolism Control
Acronym: OLFAMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2019-01909;me19ChristCrain
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Obesity
Keywords: D-limonene; lavender oil (SLVO); Olfactory stimulation; Obesity; glucose metabolism
MeSH Terms: conditions — Obesity | interventions — Limonene

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental1 (Active Comparator): During the Cross-Over study, patients will be randomly assigned to one of the arms:
  Treatment sequence: Placebo at the baseline visit, olfactory Stimulation with D-Limonene at visit 2 and olfactory Stimulation with lavender oil (SLVO) at visit 3
  Interventions: Other: D-Limonene; Other: SLVO
- Experimental2 (Active Comparator): During the Cross-Over study, patients will be randomly assigned to one of the arms:
  Treatment sequence: Placebo at the baseline visit, olfactory Stimulation with SLVO at visit 2 and olfactory Stimulation with D-Limonene at visit 3
  Interventions: Other: D-Limonene; Other: SLVO

INTERVENTIONS:
Other: D-Limonene — Patient will put the aspUraclip®, a commercially available mini-inhalator filled for our study purpose filled with 1% D-Limonene in the nose for 15 minutes
Other: SLVO — Patient will put the aspUraclip®, a commercially available mini-inhalator filled for our study purpose filled with 1% SLVO in the nose for 15 minutes

SUMMARY:
In this preliminary short-term study it is investigated, whether a short olfactory stimulation with D-Limonene leads to an acute improvement of glucose metabolism in patients with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Obesity (BMI ≥35 kg/m2)
* Written informed consent
* Normosmia (defined by sniffin Sticks test)

Exclusion Criteria:

* Known allergy to D-Limonene, citrus fruits, citrus flavours, SLVO
* Regular smoking
* Current illicit drug abuse including daily marijuana and cannabidiol (CBD) consumption (alcohol ≤2 drinks per day allowed)
* Diabetes mellitus
* Pre-Treatment with insulin sensitizing drugs including GLP-1 analogues
* History of neurodegenerative diseases, severe head trauma
* Severe renal impairment (e.g. estimated glomerular filtration rate <30 ml/min/m2)
* Known liver cirrhosis or other severe liver impairment
* Acute upper respiratory tract infection
* Uncontrolled dysthyroidism
* Uncontrolled hypertension
* Regular use of psychopharmaceutic drugs
* Patient aims to start a new diet or exercise program during the study
* Bariatric surgery
* Pregnancy/Lactation
* Symptoms of menopause
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* Participation in an interventional study within the last 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Change of area under blood glucose curve (AUBGC) | Time Frame: baseline blood exam (timepoint 0) and further blood collections: 5, 15, 30, 60, 90 and 120 minutes after drinking a standardized mixed-meal solution
  area under the blood glucose curve (AUBGC) during a mixed-meal test after stimulation with D-Limonene compared to baseline

SECONDARY OUTCOMES:
AUBGC | Time Frame: baseline blood exam (timepoint 0) and further blood collections: 5, 15, 30, 60, 90 and 120 minutes after drinking a standardized mixed-meal solution
  AUBGC during a mixed-meal test after stimulation with SLVO compared to baseline
Visual Analogue Scale (VAS score) | Time Frame: baseline VAS score (timepoint 0) and VAS scores will be evaluated after 15, 30, 60, 90 and 120 minutes after drinking a standardized mixed-meal solution
  VAS scores on hunger, appetite, nausea, mood, and hedonics of odour and/or taste of the mixed-meal shake, where 0 equals none, and 10 the maximum of each category
Change in plasma insulin levels | Time Frame: baseline blood exam (timepoint 0) and further blood collections: 5, 15, 30, 60, 90 and 120 minutes after drinking a standardized mixed-meal solution
  Plasma insulin levels (mIU/L)
Change in plasma peak glucose levels | Time Frame: baseline blood exam (timepoint 0) and further blood collections: 5, 15, 30, 60, 90 and 120 minutes after drinking a standardized mixed-meal solution
  Plasma peak glucose levels (mmol/L)
Change in plasma levels of glucagon-like peptide 1 (GLP-1) | Time Frame: baseline blood exam (timepoint 0) and further blood collections after 5, 15, 30, 60, 90 and 120 minutes after drinking a standardized mixed-meal solution
  Plasma levels of GLP-1 (pmol/L)
Change in plasma levels of gastric inhibitory polypeptide (GIP) | Time Frame: baseline blood exam (timepoint 0) and further blood collections after 5, 15, 30, 60, 90 and 120 minutes after drinking a standardized mixed-meal solution
  Plasma levels of GIP (pmol/L)
Change in plasma levels of Ghrelin | Time Frame: baseline blood exam (timepoint 0) and further blood collections after 5, 15, 30, 60, 90 and 120 minutes after drinking a standardized mixed-meal solution
  Plasma levels of Ghrelin (pg/ml)
Change in plasma levels of Leptin | Time Frame: baseline blood exam (timepoint 0) and further blood collections after 5, 15, 30, 60, 90 and 120 minutes after drinking a standardized mixed-meal solution
  Plasma levels of Leptin (ng/ml)
Change in plasma levels of Peptide YY (PYY) | Time Frame: baseline blood exam (timepoint 0) and further blood collections after 5, 15, 30, 60, 90 and 120 minutes after drinking a standardized mixed-meal solution
  Plasma levels of PYY (pg/ml)
Change in plasma levels of Glucagon | Time Frame: baseline blood exam (timepoint 0) and further blood collections after 5, 15, 30, 60, 90 and 120 minutes after drinking a standardized mixed-meal solution
  Plasma levels of Glucagon (pmol/L)
Change in plasma Levels of Interleukin-6 | Time Frame: baseline blood exam (timepoint 0) and further blood collections after 5, 15, 30, 60, 90 and 120 minutes after drinking a standardized mixed-meal solution
  Plasma Levels of Interleukin-6 (pg/ml)
Change in plasma Levels of C-reactive protein | Time Frame: baseline blood exam (timepoint 0) and further blood collections after 5, 15, 30, 60, 90 and 120 minutes after drinking a standardized mixed-meal solution
  Plasma Levels of C-reactive protein (μg/ml)
Change in plasma levels of lipids like LDL-cholesterine, total cholesterine, triglycerides | Time Frame: baseline blood exam (timepoint 0) and further blood collections: 5, 15, 30, 60, 90 and 120 minutes after drinking a standardized mixed-meal solution
  Plasma levels of lipids (mmol/L) like LDL-cholesterine, total cholesterine, triglycerides
Change in heart rate | Blood pressure and heart rate will be measured at the following times: baseline (timepoint 0) and 30, 60, 120 minutes drinking a standardized mixed-meal solution
  Heart rate (heart beats per minute)
Change in blood pressure | Blood pressure and heart rate will be measured at the following times: baseline (timepoint 0) and 30, 60, 120 minutes drinking a standardized mixed-meal solution
  blood pressure (mm Hg)

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Timper, Dr. med, Principal Investigator — Endocrinology, Diabetology and Metabolism, University Hospital Basel
Locations (1):
- Clinic for Intensive Care Medicine, University Hospital Basel, Basel, Switzerland